CLINICAL TRIAL: NCT03079999
Title: Prospective, Randomized, Placebo-Controlled Phase II Trial of Aspirin for Vestibular Schwannomas
Brief Title: Study of Aspirin in Patients With Vestibular Schwannoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, D. Bradley Welling, MD, PhD, Walter Augustus Lecompte Distinguished Professor Harvard Department of Otolaryngology-Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-030; W81XWH-17-1-0644 (Other Grant/Funding Number: Congressionally Directed Medical Research Program)
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Vestibular Schwannoma; Acoustic Neuroma; Neurofibromatosis 2
MeSH Terms: conditions — Neuroma, Acoustic; Neurofibromatosis 2 | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: In the Randomized Treatment Phase, patients aged 12 years or older with VSs will be identified and recruited into one of two randomized groups who receive either 1) 325 mg aspirin twice daily (81 mg aspirin twice daily for pediatric patients <50 kg); or 2) a placebo. Patients will stay on aspirin/placebo as long as there is no more than 20% increase in VS volume. At tumor progression, patients will enter the Open Label Follow Up Phase. Patients who progress on placebo will receive unblinded aspirin. Patients who progress on aspirin (either blinded or unblinded) will be taken off study drug and followed. All patients will be followed for at least 3.5 years after randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Patients on the experimental arm will receive blinded aspirin. Pediatric subjects who weigh less than 110 lbs will take 81mg aspirin twice a day. All other subjects will take 325mg aspirin twice a day.
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Patients on the placebo arm will receive blinded placebo and take it twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Twice daily aspirin
  Other Names: Zoprin; Durlaza; Bayer
  Arms: Aspirin
Drug: Placebo — Twice daily placebo
  Arms: Placebo

SUMMARY:
This is a phase II prospective, randomized, double-blind, longitudinal study evaluating whether the administration of aspirin can delay or slow tumor growth and maintain or improve hearing in VS patients.

DETAILED DESCRIPTION:
This is a phase II prospective, randomized, double-blind, longitudinal study evaluating whether the administration of aspirin can delay or slow tumor growth and maintain or improve hearing in VS patients. In the Randomized Treatment Phase, patients aged 12 years or older with VSs will be identified and recruited into one of two randomized groups who receive either 1) 325 mg aspirin twice daily (81 mg aspirin twice daily for pediatric patients <50 kg); or 2) a placebo. Patients will stay on aspirin/placebo as long as there is no more than 20% increase in VS volume. At tumor progression, patients will enter the Open Label Follow Up Phase. Patients who progress on placebo will be given the option to receive unblinded aspirin and will be followed until further progression, receiving a definitive treatment (e.g, surgery or radiation), or 42 months post-baseline, whichever occurs first. Patients who progress on aspirin (either blinded or unblinded) will be taken off study drug and followed until they receive a definitive treatment (e.g., surgery or radiation) or reach 42 months post-baseline, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic diagnosis of vestibular schwannoma (NF2-associated or sporadic).
* Age≥12 years.
* Ability to provide informed consent.Pediatric patients must provide assent in addition to their parents'/guardians' consent. Adult patients who cannot consent for themselves will not be eligible to participate in this study.
* Ability to swallow tablets.

Exclusion Criteria:

* Inability to perform volumetric measurements of vestibular schwannoma(s).
* Inability to tolerate MRI with contrast.
* Daily use of aspirin within the last two months. Occasional use of aspirin for pain relief is not exclusionary.
* Known allergy to aspirin.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of aspirin.
* Pregnant or lactating women.
* Patients with serious medical illnesses (e.g. severe asthma) that in the option of the investigator could prevent participation in the trial.
* Active bleeding diathesis.
* Hydrocephalus from brainstem compression.
* Febrile illness or flu-like illness in children and adolescents less than 18 years of age.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Progression, or around 3.5 years
  Progression Free Survival (PFS) is the length of time from start of study treatment to tumor growth of more than 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantina Stankovic, MD, PhD, Principal Investigator — Stanford University; D. Bradley Welling, MD, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (5):
- United States (5):
  - Stanford Otolaryngology/HNS, Stanford, California
  - University of Miami, Miami, Florida
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No